CLINICAL TRIAL: NCT01395693
Title: Assessment of the Performance of the Salt Lake Mask System as a Patient Interface in the Provision of Positive Airway Pressure (PAP) Therapy
Brief Title: Performance of the Salt Lake Mask System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MA200611
Record Dates: First submitted 2011-06-29; First posted 2011-07-15 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Salt Lake mask system (Experimental)
  Interventions: Device: Salt Lake mask system

INTERVENTIONS:
Device: Salt Lake mask system — Study participants will Salt Lake mask system for 1 week in place of their current mask system.
  Other Names: Salt Lake

SUMMARY:
Assessment of the performance of the Salt Lake mask system acting as a patient interface in the provision of PAP therapy. This study will assess the suitability of this mask system in its current form for use.

DETAILED DESCRIPTION:
Sleep-disordered breathing (SDB) is a significant direct cause of morbidity and mortality, as well as being a significant indirect cause of morbidity and mortality impacting greatly upon health and quality of life when left untreated. Positive Airway Pressure (PAP) therapy is an effective and proven form of medical treatment for many types of SDB.

In order for PAP therapy to be effective, patient interfaces(masks) need to be both effective in their delivery of this treatment and accepted by prospective and current patients for use. This study will investigate the ability of the Salt Lake mask system to act effectively as a patient interface in PAP therapy, and its ability to be accepted by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients using the Swift FX mask system
* Patients who can trial the mask for 7 nights
* Patients who have used PAP therapy for a minimum of 6 months.

Exclusion Criteria:

* Patients not willing to give written informed consent
* Patients who can not read and comprehend English
* Patients using an inappropriate mask system
* Patients using Bilevel flow generators
* Patients who are pregnant
* Patients who are unable to comply with the protocol
* Patients who have used PAP therapy for less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Subjectively Assessed Levels of Seal, Comfort, Stability and Overall Performance. | 1 week
  Participants in the study will complete a subjective assessment of the levels of seal, comfort, stability and overall Performance of Salt Lake Mask System in use.

SECONDARY OUTCOMES:
Subjective Assessments of Ease and Intuitiveness in Assembly and Disassembly | 1 week
  Participants in the study will subjectively assess the ease and intuitiveness of specific common assembly/diosassembly tasks related to the Salt Lake mask system.
Subjectively Assessed Levels of Skin Markings | 1 week
  Participants in the study will subjectively assess the levels of Skin Markings experienced as a direct result of use of the Salt Lake mask system.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, Principal Investigator — ResMed
Locations (1):
- ResMed Ltd, Sydney, New South Wales, Australia